CLINICAL TRIAL: NCT06632223
Title: The Effect of Sensory Motor Training on Foot Weight Distribution and Postural Stability in Patients With Foot Burn
Brief Title: Sensory Motor Training on Foot Weight Distribution in Patients With Foot Burn
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shaimaa Mohamed Ahmed Elsayeh (Other)
Responsible Party: Sponsor-Investigator, Shaimaa Mohamed Ahmed Elsayeh, Assistant Professor of Physical Therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005257
Record Dates: First submitted 2024-09-28; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Burn; Postural Stability
Keywords: Sensory motor training; Foot weight distribution; Postural stability; Foot burn
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sensory-motor training group (Experimental): This group will include 35 patients with foot burns. Patients will receive sensorimotor training exercise in addition to a traditional physical therapy program in the form of stretching exercises, strengthening exercises and scar management. Exercises will be applied for 3 times a week for 8 consecutive weeks.
  Interventions: Other: Sensory motor training; Other: Traditional physical therapy
- Traditional physical therapy group (Active Comparator): This group will include 35 patients with foot burns. Patients will receive the traditional physical therapy program only in the form of stretching exercises, strengthening exercises and scar management. Exercises will be applied for 3 times a week for 8 consecutive weeks.
  Interventions: Other: Traditional physical therapy

INTERVENTIONS:
Other: Sensory motor training — Each session will be composed of 10 minutes of warm-up, followed by 50-60 minutes of sensory motor exercises, followed by 5-10 minutes of cool down.
  Arms: Sensory-motor training group
Other: Traditional physical therapy — traditional physical therapy program in form of stretching exercises, strengthening exercises, scar management, and gait training

SUMMARY:
The purpose of the current study is to investigate the effect sensory motor training on foot weight distribution and postural stability in patients with foot burn.

DETAILED DESCRIPTION:
Pain, contractures, scars, altered sensations, muscle weakness, and postural balance impairment are potential complications of foot burn that negatively influence a person's ability to function normally and correlate with gait abnormalities like reduced step height and length, along with slower gait speed. These gait disturbances pose significant challenges for burn patients, affecting their mobility and overall quality of life. So, this study aims to understanding how sensory motor training can improve balance, gait, and overall functional mobility is essential for guiding the development of evidence-based rehabilitation protocols tailored to the unique needs of this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients will suffer from foot "planter surface" second degree thermal burn (Partial thickness).
* Patients who have undergone skin grafting and those who have not undergone skin grafting are both eligible for inclusion in the study.
* Patients will begin the training program after complete wound healing.
* Patients will be given their informed consent.

Exclusion Criteria:

* Patients who had an open wound at or near treatment site.
* Patients who had chemical or electrical burn.
* Patients with specific conditions such as musculoskeletal impairments impacting independent walking (e.g., strokes, severe arthritis).
* Uncontrolled cardiovascular or pulmonary diseases.
* Patients with neurological, psychiatric illness, severe behavior or cognitive disorders.
* Metabolic or vascular disease with a neurological component such as diabetes.
* Patients with hearing problems, individuals with otitis media, and patients experiencing nystagmus and visual problems.
* Malignant conditions.
* Uncooperative patients.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The Pedoscan system | "At baseline and after 8 weeks of intervention"
  It will be used to assess the foot weight distribution. Under the guidance of the evaluator, the subjects will stand with bare feet upon a part marked on the platform with eyes closed.
The biodex balance system | "At baseline and after 8 weeks of intervention"
  It will be used to assess the postural stability during assessment; participants will stand comfortably on the platform barefoot, with arms at their sides, for 30 seconds.

SECONDARY OUTCOMES:
The Brief Burn Specific Health Scale-Brief | "At baseline and after 8 weeks of intervention"
  Its Arabic version will be used to assess the quality of life. The Burn Specific Health Scale-Brief consists of 40 items covering nine domains related to health-related quality of life (HRQL): simple abilities, heat sensitivity, hand function, treatment regimens, work, body image, affect, interpersonal relationships, and sexuality. Responses to each item are scored on a five-point scale ranging from 0 (extremely) to 4 (not at all). Mean scores per domain are assessed, and high scores indicate a good perceived health status

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Cairo University, Egypt., Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No